CLINICAL TRIAL: NCT03194464
Title: Neural Mechanisms Mediating Interlimb Transfer Following Stroke
Brief Title: Fatiguing Arm Exercise Following Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N1759-P
Record Dates: First submitted 2016-10-14; First posted 2017-06-21 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Stroke
Keywords: hemiparesis
MeSH Terms: conditions — Stroke; Paresis | interventions — Hand Strength

STUDY DESIGN:
Intervention Model Description: Prospective, repeated measures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Task-failure, Extended Session (Experimental): Repeated sub-maximal gripping exercise with the less affected hand to task-failure - followed by repeated measurements (5) during recovery period
  Interventions: Other: submaximal exercise (grip)

INTERVENTIONS:
Other: submaximal exercise (grip) — participants perform repeated gripping with visual feedback to task failure

SUMMARY:
This study investigates the effects of sub-maximal exercise to task-failure (e.g., fatigue) with the less involved, or so-called non-paretic hand, in people who have experienced a stroke. In previous work the investigators found that non-paretic hand exercise to task-failure increased excitability of the motor cortex in the more involved hemisphere and produced behavioral improvements in the unexercised paretic hand. Importantly, the magnitude of increased brain excitability is greater than what has been observed following brain stimulation with either repetitive transcranial magnetic stimulation (TMS) or transcranial direct current stimulation (tDCS) and lasts longer. This approach could be implemented in the clinical setting and could be accessible to a greater number of people than brain stimulation. The investigators' goals in the current study are to: repeat previous findings in a different group of participants and investigate the neural mechanisms that produce brain and behavioral facilitation in order to inform development of this approach for clinical implementation.

DETAILED DESCRIPTION:
The long-term goal is to restore upper extremity (UE) motor function following stroke. The overall objective of this proposal is to improve the investigators' understanding of neural mechanisms contributing to inter-limb and inter-hemispheric transfer following non-paretic limb exercise to task failure. The investigators will use transcranial magnetic stimulation to probe acute adaptations in cortical excitability, intracortical and inter-hemispheric circuits that accompany behavioral facilitation of the paretic hand.

The work proposed in this two year project will enable the investigators to obtain three data elements critical to complete the working hypothesis:

1. . Changes in intracortical and interhemispheric inhibition in both hemispheres following non-paretic limb exercise to task-failure.
2. . Behavioral effects using a motor task involving manipulation and dexterity.
3. . Determine the persistence and consistency of neural and behavioral facilitation.

ELIGIBILITY:
Inclusion Criteria:

* individuals at least 6 months post-stroke in the cortical or sub-cortical distribution with residual upper-extremity hemiparesis
* Non-Veteran Participants are eligible

Exclusion Criteria:

* multiple strokes
* strokes in both hemispheres
* brainstem/medullary/cerebellar stroke
* seizure disorder
* metal implants in head or neck
* pacemaker or other implanted device
* inability to produce any measurable grip force

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolynn Patten, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants identified by the VA Brain Rehabilitation Research Center (BRRC) screening and recruitment core enrolled between 2/1/2016 - 5/21/2018.
Groups:
- Task-Failure, Extended Session: individuals with upper-extremity impairment resulting from stroke, enrolled six or more months following stroke performed submaximal exercise (grip): participants performed submaximal gripping with the non-paretic hand to task failure, guided by visual feedback. Recovery was monitored for an extended period of 3:45 following task-failure.
Period: Overall Study
Arm/Group | Task-Failure, Extended Session
Started | 15
Completed | 13
Not Completed | 2
Not completed — data not usable | 2

BASELINE CHARACTERISTICS:
Population: No differences from inclusion criteria. As noted, data were not usable from 2 participants, thus only 13 data sets were analyzed.
Groups:
- Task-failure, Extended Session: Exercise to fatigue followed by repeated monitoring of recovery until 3:45 after.
Arm/Group | Task-failure, Extended Session
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years]
  Extended Session | 61.1 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Upper-extremity Fugl-Meyer Motor Assessment [Mean (Standard Deviation); unit: units on a scale] — The Fugl-Meyer Motor Assessment is a widely-used validated measure of motor impairment for individuals post-stroke. The upper-extremity component totals 66 points. Higher scores reflect less impairment/less severe hemiparesis, although 66 points is not equivalent to "normal" or scores achieved by non-disabled individuals. Lower scores reflect greater impairment/more severe hemiparesis.
  units on a scale | 54.6 (13.2)
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units on a scale] — The Montreal Cognitive Assessment (MoCA) is a cognitive screening test designed to detect mild cognitive impairment and more serious cognitive disorders such as dementia. The scale ranges from 0 - 30 points; scores 26 and greater are considered normal.
  units on a scale | 27.0 (1.96)
Center for Epidemiologic Studies - Depression Scale [Mean (Standard Deviation); unit: units on a scale] — The Center for Epidemiologic Studies - Depression Scale (CES-D) was designed to measure self-reported symptoms of depression experienced in the prior week. Scores range from zero -to - 60 with higher scores representing greater incidence of symptomatology.
  units on a scale | 9.0 (9.3)
Fatigue Severity Scale [Mean (Standard Deviation); unit: units on a scale] — The Fatigue Severity Scale (FSS) is a patient-reported outcome evaluating the impact of fatigue on the individual designed to differentiate fatigue from clinical depression. Scores range from 0 - to - 7. People with depression alone score ~4.5, while people with fatigue related to an underlying neurological condition score ~6.5.
  units on a scale | 3.95 (1.58)

OUTCOME MEASURES:

1. Primary Outcome: Short Intracortical Inhibition (SICI)
Description: SICI is a neurophysiologic measure of intra-cortical inhibition, obtained using transcranial magnetic stimulation (TMS) measured here in the ipsilesional hemisphere (IH) at each point to determine how it is modulated in response to task-failure. SICI is quantified as a ratio where values <1 reflect inhibition and >1 disinhibition or relative excitation. In health, SICI is ~0.5. Thus if SICI = 0.8, while <1 it would indicate less inhibition than expected in health. Transient change in SICI from 0.8 to 1.1 over the course of this experimental paradigm would reflect a period of relative excitation in response to the exercise paradigm.
Time Frame: baseline, post task-failure (minutes to an hour), every 45 min up to 3.5 hours post-task-failure (7 points total)
Population: Only 13/15 data sets were usable for reasons explained elsewhere in the record. Thus, while 15 individuals were enrolled, we were able to analyze only 13 of these individuals' data.
Measure: Mean (Standard Error); unit: SICI ratio
Groups:
- Task-Failure, Extended Session: individuals with upper-extremity impairment following stroke
  submaximal exercise (grip): participants perform repeated gripping with visual feedback to task failure
Arm/Group | Task-Failure, Extended Session
Number analyzed (Participants) | 13
SICI ratio
  Baseline | 0.83 (0.07)
  0 min post-task-failure | 1.14 (0.15)
  45 min post-task-failure | 0.89 (0.11)
  90 min post-task-failure | 0.88 (0.05)
  135 min post-task-failure | 0.82 (0.06)
  180 min post-task-failure | 0.87 (0.06)
  225 min post-task-failure | 0.81 (0.06)
Statistical Analysis 1: Comparison: Task-Failure, Extended Session; We performed repeated measures analysis of variance (RM-ANOVA) to determine if intracortical inhibition, as measured by SICI, in the ipsilesional hemisphere was altered by less affected hand exercise to task-failure and to determine the time course and recovery of this effect; Test type: Other; p = 0.15, ANOVA — The a priori threshold for statistical significance was established at p <.05 (non-adjusted)

2. Primary Outcome: SICI Ratio
Description: as for outcome 1
Time Frame: Baseline, pre-exercise of 8 repeated sessions
Population: Only 10/12 data sets analyzed because it was possible to induce SICI in only 10 individuals.
Measure: Mean (Standard Deviation); unit: SICI ratio
Groups:
- Task-failure, Repeated Sessions: Individuals with upper-extremity motor impairment following stroke. Performed 8 repeated sessions of exercise to task-failure (2x per week x 4 weeks)
Arm/Group | Task-failure, Repeated Sessions
Number analyzed (Participants) | 10
SICI ratio
  Session1 | 0.89 (0.25)
  Session2 | 0.85 (0.14)
  Session3 | 0.93 (0.29)
  Session4 | 0.80 (0.29)
  Session5 | 0.78 (0.28)
  Session6 | 0.77 (0.37)
  Session7 | 0.88 (0.25)
  Session8 | 0.83 (0.31)
Statistical Analysis 1: Comparison: Task-failure, Repeated Sessions; We performed repeated measures analysis of variance (RM-ANOVA) to determine if intracortical inhibition, as measured by SICI, in the ipsilesional hemisphere was altered by repeated sessions of less affected hand exercise to task-failure. Pre-exercise SICI was compared between Session1 and Session8; Test type: Superiority; p = .83, ANOVA — Statistical Significance established as p <.05; Repeated-Measures ANOVA

3. Other Pre Specified Outcome: Box and Blocks Test (BBT)
Description: The BBT measures motor function/dexterity, scored as the number of blocks transferred in 1 minute. Here function of the paretic hand was measured at each time point: baseline, post-task failure, 45min post, 90min post, 135min post, 180min post, 225min post-task failure to determine the change in paretic hand BBT performance following exercise to task-failure. Scores are numeric ranging from 0 (no blocks transferred) to whatever the participant is able to achieve. Healthy age-matched adults without motor disability score in the range of 60 (+/- 10) blocks transferred in 1 minute.
Time Frame: baseline, post task-failure (requires variable timeline from minutes to an hour), every 45 min up to 3.5 hours post-task-failure (7 points total)
Population: The Box and Blocks test (BBT) is an accepted measure of motor function/dexterity. Score reflect the number of 1" blocks moved from one half of a divided box to the other in 1 minute. Higher numbers indicate better performance.
  Only 13/15 data sets were analyzed because other data sets were not usable.
Measure: Mean (Standard Error); unit: blocks
Groups:
- Task-failure, Extended Session: individuals with upper-extremity impairment resulting from stroke, enrolled six or more months following stroke
  submaximal exercise (grip): participants performed repeated gripping with the non-paretic hand to task failure. Visual feedback was provided.
Arm/Group | Task-failure, Extended Session
Number analyzed (Participants) | 13
blocks
  Baseline | 25.4 (3.6)
  0 min post-task-failure | 25.5 (3.2)
  45 min post-task-failure | 25.0 (3.3)
  90 min post-task-failure | 26.1 (3.4)
  135 min post-task-failure | 26.7 (3.6)
  180 min post-task-failure | 25.7 (3.6)
  225 min post-task-failure | 26.9 (3.7)
Statistical Analysis 1: Comparison: Task-failure, Extended Session; RM-ANOVA; Test type: Other; p = 0.204, ANOVA

4. Other Pre Specified Outcome: Box and Blocks Test (BBT)
Description: The BBT measures motor function/dexterity, scored as the number of blocks transferred in 1 minute. Here function of the paretic hand was measured prior to exercise at each of 8 repeated sessions conducted twice weekly for 4 weeks to determine the change in paretic hand BBT performance following repeated sessions of exercise to task-failure. Scores are numeric ranging from 0 (no blocks transferred) to whatever the participant is able to achieve. Healthy age-matched adults without motor disability score in the range of 60 (+/- 10) blocks transferred in 1 minute.
Time Frame: baseline, pre-exercise of 8 repeated sessions
Population: BBT data were obtained in all 12 individuals at each of 8 sessions.
Measure: Mean (Standard Deviation); unit: blocks
Arm/Group | Task-failure, Repeated Sessions
Number analyzed (Participants) | 12
blocks
  Session1 | 23.2 (12.8)
  Session2 | 23.5 (13.2)
  Session3 | 26.8 (11.5)
  Session4 | 28.5 (11.9)
  Session5 | 27.4 (12.7)
  Session6 | 29.8 (10.9)
  Session7 | 29.7 (11.8)
  Session8 | 29.3 (11.9)
Statistical Analysis 1: Comparison: Task-failure, Repeated Sessions; We performed repeated measures analysis of variance (RM-ANOVA) to determine if motor dexterity, as measured by the BBT, was improved by repeated sessions of non-paretic hand exercise to task-failure. BBT performance was compared between Session1 and Session8; Test type: Superiority; p = .004, ANOVA — statistical significance was established a priori at p <.05; repeated measures ANOVA comparing Session8 vs. Session1 performance

ADVERSE EVENTS:
Time Frame: Study Duration, 2 years.
Description: This was a low risk study of exercise.
Arm/Group | Task-failure, Extended Session
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
This was designed and intended as a small, pilot study to establish feasibility, refine methods, and generate preliminary data that could motivate sample size projections for future study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT03194464/Prot_SAP_000.pdf